CLINICAL TRIAL: NCT00117702
Title: Prophylaxis of the Graft-Versus-Host-Disease in Patients After Allogeneic Stem Cell Transplantation With a Combination of Tacrolimus and Everolimus
Brief Title: Prevention of the Graft-Versus-Host-Disease in Patients After Stem Cell Transplantation With Tacrolimus and Everolimus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: safety reasons
Sponsor: Technische Universität Dresden (Other)
Responsible Party: TUD, Technical University Dresden
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30; 2005-000161-19 (EudraCT Nr.)
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Graft vs Host Disease
Keywords: GvHD; Tacrolimus; Everolimus; Stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tacrolimus — day 0-100, then taper
  Other Names: Prograf
Drug: Everolimus — day 0-56
  Other Names: Certican

SUMMARY:
The purpose of this pilot study is to provide preliminary data about the efficacy and the safety of the combination of tacrolimus with everolimus in the prophylaxis of the graft-versus-host-disease (GvHD) in patients after allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
The allogeneic stem cell transplantation is a successful therapeutic approach in the treatment of a number of hematologic diseases. Nevertheless, it is associated with substantial risks and complications. A major life-threatening complication that occurs in the post transplantation period is the graft versus host disease, especially its severe forms (Grade III and Grade IV). For this reason, a combined immunosuppressive therapy is standard in patients after a stem cell transplantation. In this regard, the combination between cyclosporin A and methotrexate in the prevention of GvHD has been particularly successful. However, the incidence rate of GvHD and consequent mortality are still fairly high. Besides, the therapy itself is accompanied by serious side effects. Therefore, there is a need for a more efficient, less toxic, combined immunosuppressive therapy. The purpose of this pilot study is to test a new combination of immunosuppressives (tacrolimus and everolimus) for the prevention of GvHD after an allogeneic stem cell transplantation. Tacrolimus is a macrolide immunosuppressant that acts as a calcineurin inhibitor, thereby preventing the activation and proliferation of the T-lymphocytes. Everolimus is a semisynthetic macrocyclic lactone that inhibits the activity of a key protein involved in the regulation of the cell cycle, the so called m-TOR protein. Both medicaments act complementary and potently inhibit the proliferation of immune cells. Previous studies have shown that the combination of tacrolimus with everolimus decreases significantly the rejection rate after solid organ transplantation and this combination is generally well tolerated.

This study is designed as a prospective, single-center, non-randomized, open-label non-controlled pilot study. Study related visits are scheduled to take place at regular time intervals and the patients will be followed up to one year after the stem cell transplantation. The study is designed and will be conducted in accordance with the ICH-GCP guidelines and the respective national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 70 years of age
* Planned allogeneic stem cell transplantation either from a related or an unrelated donor
* Written informed consent

Exclusion Criteria:

* Previous stem cell transplantation
* Use of antibody Campath (anti CD-52) or ATG during the conditioning
* In vitro T-cell depleted graft
* Known hypersensitivity to everolimus or other constituents of the study medication
* Symptomatic infectious disease
* Hepatic disease (ASAT > 2 x ULN)
* Renal insufficiency (creatinine > 2 x ULN)
* HIV infection
* Life expectancy < 3 months
* Severe lung disease (FEV1 < 50% of the normal value)
* Severe psychiatric disorder
* Subjects unlikely to comply with the requirements of the protocol
* Known or current alcohol, medication or drug abuse
* Pregnancy or lactation
* Women of child-bearing potential without reliable contraception unless they meet the following criteria: postmenopausal (12 months of natural amenorrhea);postoperation status (6 weeks after surgical bilateral oophorectomy with or without hysterectomy);use of highly effective birth control method (defined as one which results in a low failure rate i.e. less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or vasectomized partner)
* Men that do not use one of the following methods for prevention of conception:sexual abstinence; condom; vasectomy
* Participation of the subject in another clinical trial within the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GvHD grade III and IV within the first 100 days after the stem cell transplantation | first 100 days

SECONDARY OUTCOMES:
Safety (evaluated after Common Terminology Criteria for Adverse Events [CTCAE] v 3.0) | within 100 days after Tx
Hypersensitivity reactions | within 56 days after Tx
Thrombotic thrombocytopenic purpura | within 56 days after Tx
Hyperlipidemia | within 56 days after Tx
Total and relapse-free survival rate one year after the stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, Principal Investigator — University Clinic Carl Gustav Carus Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, University Clinic Carl Gustav Carus, Dresden, Germany

REFERENCES:
- [Background] Antin JH, Kim HT, Cutler C, Ho VT, Lee SJ, Miklos DB, Hochberg EP, Wu CJ, Alyea EP, Soiffer RJ. Sirolimus, tacrolimus, and low-dose methotrexate for graft-versus-host disease prophylaxis in mismatched related donor or unrelated donor transplantation. Blood. 2003 Sep 1;102(5):1601-5. doi: 10.1182/blood-2003-02-0489. Epub 2003 May 1. PMID 12730113
- [Background] Barten MJ, Streit F, Boeger M, Dhein S, Tarnok A, Shipkova M, Armstrong VW, Mohr FW, Oellerich M, Gummert JF. Synergistic effects of sirolimus with cyclosporine and tacrolimus: analysis of immunosuppression on lymphocyte proliferation and activation in rat whole blood. Transplantation. 2004 Apr 27;77(8):1154-62. doi: 10.1097/01.tp.0000120391.42712.e8. PMID 15114077
- [Background] Bornhauser M, Schuler U, Porksen G, Naumann R, Geissler G, Thiede C, Schwerdtfeger R, Ehninger G, Thiede HM. Mycophenolate mofetil and cyclosporine as graft-versus-host disease prophylaxis after allogeneic blood stem cell transplantation. Transplantation. 1999 Feb 27;67(4):499-504. doi: 10.1097/00007890-199902270-00001. PMID 10071016
- [Background] Cutler C, Kim HT, Hochberg E, Ho V, Alyea E, Lee SJ, Fisher DC, Miklos D, Levin J, Sonis S, Soiffer RJ, Antin JH. Sirolimus and tacrolimus without methotrexate as graft-versus-host disease prophylaxis after matched related donor peripheral blood stem cell transplantation. Biol Blood Marrow Transplant. 2004 May;10(5):328-36. doi: 10.1016/j.bbmt.2003.12.305. PMID 15111932
- [Background] Eisen HJ, Tuzcu EM, Dorent R, Kobashigawa J, Mancini D, Valantine-von Kaeppler HA, Starling RC, Sorensen K, Hummel M, Lind JM, Abeywickrama KH, Bernhardt P; RAD B253 Study Group. Everolimus for the prevention of allograft rejection and vasculopathy in cardiac-transplant recipients. N Engl J Med. 2003 Aug 28;349(9):847-58. doi: 10.1056/NEJMoa022171. PMID 12944570
- [Background] Gratwohl A, Brand R, Apperley J, Biezen Av Av, Bandini G, Devergie A, Schattenberg A, Frassoni F, Guglielmi C, Iacobelli S, Michallet M, Kolb HJ, Ruutu T, Niederwieser D; Chronic Leukemia Working Party of the European Group for Blood and Marrow Transplantation (CLWP-EBMT). Graft-versus-host disease and outcome in HLA-identical sibling transplantations for chronic myeloid leukemia. Blood. 2002 Dec 1;100(12):3877-86. doi: 10.1182/blood.V100.12.3877. PMID 12433695
- [Background] Hackstein H, Taner T, Zahorchak AF, Morelli AE, Logar AJ, Gessner A, Thomson AW. Rapamycin inhibits IL-4--induced dendritic cell maturation in vitro and dendritic cell mobilization and function in vivo. Blood. 2003 Jun 1;101(11):4457-63. doi: 10.1182/blood-2002-11-3370. Epub 2003 Jan 16. PMID 12531798
- [Background] Hoyer PF, Ettenger R, Kovarik JM, Webb NJ, Lemire J, Mentser M, Mahan J, Loirat C, Niaudet P, VanDamme-Lombaerts R, Offner G, Wehr S, Moeller V, Mayer H; Everolimus Pediatric Study Group. Everolimus in pediatric de nova renal transplant patients. Transplantation. 2003 Jun 27;75(12):2082-5. doi: 10.1097/01.TP.0000070139.63068.54. PMID 12829916
- [Background] Kovarik JM. Everolimus: a proliferation signal inhibitor targeting primary causes of allograft dysfunction. Drugs Today (Barc). 2004 Feb;40(2):101-9. doi: 10.1358/dot.2004.40.2.799422. PMID 15045032
- [Background] Kovarik JM, Kaplan B, Silva HT, Kahan BD, Dantal J, McMahon L, Berthier S, Hsu CH, Rordorf C. Pharmacokinetics of an everolimus-cyclosporine immunosuppressive regimen over the first 6 months after kidney transplantation. Am J Transplant. 2003 May;3(5):606-13. doi: 10.1034/j.1600-6143.2003.00107.x. PMID 12752317
- [Background] MacDonald AS. Rapamycin in combination with cyclosporine or tacrolimus in liver, pancreas, and kidney transplantation. Transplant Proc. 2003 May;35(3 Suppl):201S-208S. doi: 10.1016/s0041-1345(03)00231-8. PMID 12742497
- [Background] Monti P, Mercalli A, Leone BE, Valerio DC, Allavena P, Piemonti L. Rapamycin impairs antigen uptake of human dendritic cells. Transplantation. 2003 Jan 15;75(1):137-45. doi: 10.1097/00007890-200301150-00025. PMID 12544886
- [Background] Nash RA, Antin JH, Karanes C, Fay JW, Avalos BR, Yeager AM, Przepiorka D, Davies S, Petersen FB, Bartels P, Buell D, Fitzsimmons W, Anasetti C, Storb R, Ratanatharathorn V. Phase 3 study comparing methotrexate and tacrolimus with methotrexate and cyclosporine for prophylaxis of acute graft-versus-host disease after marrow transplantation from unrelated donors. Blood. 2000 Sep 15;96(6):2062-8. PMID 10979948
- [Background] Panwalkar A, Verstovsek S, Giles FJ. Mammalian target of rapamycin inhibition as therapy for hematologic malignancies. Cancer. 2004 Feb 15;100(4):657-66. doi: 10.1002/cncr.20026. PMID 14770419
- [Background] Qi S, Xu D, Peng J, Vu MD, Wu J, Bekersky I, Fitzsimmons WE, Peets J, Sehgal S, Daloze P, Chen H. Effect of tacrolimus (FK506) and sirolimus (rapamycin) mono- and combination therapy in prolongation of renal allograft survival in the monkey. Transplantation. 2000 Apr 15;69(7):1275-83. doi: 10.1097/00007890-200004150-00012. PMID 10798741
- [Background] Storb R, Deeg HJ, Whitehead J, Appelbaum F, Beatty P, Bensinger W, Buckner CD, Clift R, Doney K, Farewell V, et al. Methotrexate and cyclosporine compared with cyclosporine alone for prophylaxis of acute graft versus host disease after marrow transplantation for leukemia. N Engl J Med. 1986 Mar 20;314(12):729-35. doi: 10.1056/NEJM198603203141201. PMID 3513012
- [Background] Sullivan KM, Anasetti C, Horowitz M, Rowlings PA, Petersdorf EW, Martin PJ, Clift RA, Walters MC, Gooley T, Sierra J, Anderson JE, Bjerke J, Siadak M, Flowers ME, Nash RA, Sanders JE, Appelbaum FR, Storb R, Hansen JA. Unrelated and HLA-nonidentical related donor marrow transplantation for thalassemia and leukemia. A combined report from the Seattle Marrow Transplant Team and the International Bone Marrow Transplant Registry. Ann N Y Acad Sci. 1998 Jun 30;850:312-24. doi: 10.1111/j.1749-6632.1998.tb10488.x. PMID 9668553
- [Background] Sullivan KM, Weiden PL, Storb R, Witherspoon RP, Fefer A, Fisher L, Buckner CD, Anasetti C, Appelbaum FR, Badger C, et al. Influence of acute and chronic graft-versus-host disease on relapse and survival after bone marrow transplantation from HLA-identical siblings as treatment of acute and chronic leukemia. Blood. 1989 May 1;73(6):1720-8. PMID 2653460
- [Background] Vu MD, Qi S, Xu D, Wu J, Fitzsimmons WE, Sehgal SN, Dumont L, Busque S, Daloze P, Chen H. Tacrolimus (FK506) and sirolimus (rapamycin) in combination are not antagonistic but produce extended graft survival in cardiac transplantation in the rat. Transplantation. 1997 Dec 27;64(12):1853-6. doi: 10.1097/00007890-199712270-00039. PMID 9422432
- [Background] Woltman AM, van der Kooij SW, Coffer PJ, Offringa R, Daha MR, van Kooten C. Rapamycin specifically interferes with GM-CSF signaling in human dendritic cells, leading to apoptosis via increased p27KIP1 expression. Blood. 2003 Feb 15;101(4):1439-45. doi: 10.1182/blood-2002-06-1688. Epub 2002 Sep 26. PMID 12393532
- [Background] Xu Q, Simpson SE, Scialla TJ, Bagg A, Carroll M. Survival of acute myeloid leukemia cells requires PI3 kinase activation. Blood. 2003 Aug 1;102(3):972-80. doi: 10.1182/blood-2002-11-3429. Epub 2003 Apr 17. PMID 12702506